CLINICAL TRIAL: NCT02872155
Title: Comparative Study of the Efficacy of Oral Versus Intravenous Hydration as a Preventive Measure of Contrast-induced Nephropathy (CIN) in Patients
Brief Title: Comparative Study of the Efficacy of Oral Versus Intravenous Hydration as a Preventive Measure of Contrast-induced Nephropathy (CIN) in Patients With Renal Insufficiency (RI) Grade III Under Study Conducting Computed Tomography (CT)
Acronym: NICIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: David Garcia Cinca (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor-Investigator, David Garcia Cinca, Clinical Research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NICIR
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Renal Insufficiency
Keywords: contrast-induced nephropathy; renal insufficiency; computed tomography
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral hydratation (Experimental)
  Interventions: Other: Oral hydratation
- Endovenous hydratation (Active Comparator)
  Interventions: Drug: Bicarbonate endovenous hydratation; Drug: Saline endovenous hydratation

INTERVENTIONS:
Other: Oral hydratation — 500 mL of water two hours before computed tomography and 2000 milliliters 24 hours after performing computed tomography
  Arms: Oral hydratation
Drug: Bicarbonate endovenous hydratation — Intravenous hydration: sodium (1.6 molar) Bicarbonate 3 mL / kg / h starting one hour before the computed tomography and sodium bicarbonate (1/6 M) 1 mL / kg / h during the hour after computed tomography.
  Arms: Endovenous hydratation
Drug: Saline endovenous hydratation — If there is contraindication for administration of bicarbonate the pattern of intravenous hydration is performed with saline solution: 3 ml / kg / h for 1 hour before the procedure and normal saline 1 mL / kg / hour for hour after computed tomography.
  Arms: Endovenous hydratation

SUMMARY:
This study evaluates if oral hydratation is as effective as endovenous hydratation in the prophylaxis of contrast-induced nephropathy in patients renal insufficiency grade III under study conducting contrasted computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over 18 years
* Candidates for a study with computed tomography and intravenous contrast
* A glomerular filtration rate between 30 and 45 mL / min including both determinations
* They have signed the written informed consent after being informed of the objectives and the nature of the case or be unable to have the authorization or agreement of its

Exclusion Criteria:

* refuse to participate in the study
* pregnancy or lactation
* Other risk factors for Contrast Induced Nephropathy: diabetes mellitus type I, have an age of 75 years or above, heart failure (defined by a scale New York Heart Association 3 or 4), hypotension (defined as systolic blood pressure <100), being treated with nephrotoxic medications.
* Any disease or a history that, in the investigator's opinion, could confound the results of the study or pose an additional risk to patient treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Proportion of contrast induced nephropathy | 48-72 hours after the completion of the computed tomography
  Contrast induced nephropathy defined as a creatinine increase> 0.5 mg
  / dl comparing the initial blood test to the blood test performed after 48-72 hours to the completion of the computed tomography

SECONDARY OUTCOMES:
Need for hemodialysis | 15 days
  Need for hemodialysis for one month after completion of the computed tomography, among patients who have undergone oral or intravenous hydration
Reversibility of contrast induced nephropathy | 15 days
  Defined as no increase in creatinine> 0.5 mg / dl compared to the initial analysis performed
Proportion of adverse events | 15 days
  Presence of adverse events, grade 3 adverse events and serious adverse events related to the investigational products during the study follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic i Provincial de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided